CLINICAL TRIAL: NCT06084767
Title: Evaluating the Clinical Value of 68Ga-TCR-FAPI PET/CT in Patients With Various Types of Cancer
Brief Title: 68Ga-TCR-FAPI PET/CT in Patients With Various Types of Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TCR-FAPI PET/CT in cancers
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Malignant Tumor; Positron Emission Tomography; Fibroblast Activation Protein Inhibitor
Keywords: Malignant Tumor; Positron Emission Tomography; Fibroblast Activation Protein Inhibitor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: 68Ga-TCR-FAPI PET/CT was used for patients with suspected malignant tumors
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Malignant tumors (Experimental): This arm investigated the clinical value of 68Ga-TCR-FAPI PET/CT in suspected malignant tumors.
  Interventions: Diagnostic Test: 68Ga-TCR-FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-TCR-FAPI PET/CT — A dose of 3.7 MBq/kg 68Ga-TCR-FAPI will be intravenously injected and PET examination will be carried out within the specified time.

SUMMARY:
Adding targeted covalent radiopharmaceutical (TCR) moiety to fibroblast activation protein inhibitor (FAPI) can increase tumor uptake and tumor retention in pre-clinical studies. This study is an open-labeled single-arm phase II diagnostic clinical trial to explore the clinical value of 68Ga-TCR-FAPI PET/CT in suspected malignant tumor patients.

DETAILED DESCRIPTION:
TCR-FAPI can covalently bind to FAP that increase tumor uptake and tumor retention in pre-clinical studies, which elevates the ability for cancer imaging and facilitates the targeted radionuclide therapy. This study is an open-labeled single-arm phase II diagnostic clinical trial to explore the clinical value of 68Ga-TCR-FAPI PET/CT in suspected malignant tumor patients. Quantitative features (i.e., SUVmax) will be calculated to evaluate the PET images. Alternative imaging modality, including but not limited to, Ultrasound, CT, MRI, and PET/CT with other radiotracers, might be applied according to clinical needs. For patients who took surgery after multiple examination, tumor tissue and histopathology will also be obtained. For patients who underwent other treatment, treatment response of each individual lesion will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Suspected to have malignant tumors (supported by MRI and/or CT and/or tumor markers and/or pathology report), the tumor may be newly diagnosed or previously treated;
* Meet the indications for PET examination, show a clear indication and no contraindications;
* Have a performance status of score ≥ 80 on KPS scale or score 0-1 points on ECOG scale, a relatively good general situation;
* No major organ dysfunction (heart, lung, liver, kidney and other major organ include), acute or life-threatening status of infection;
* Be ≥ 18 years of age;
* Be willing and able to understand the research content and provide written informed consent/assent for the trial.

Exclusion Criteria:

* Have a history of imaging agent allergies;
* Does not meet the PET-CT scan sedation requirements, or has contraindications for PET-CT examination;
* Be pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 90 days
  The sensitivity, specificity, and accuracy of 68Ga-TCR-FAPI PET/CT to detect tumor lesions were calculated to evaluate the diagnostic efficacy.

SECONDARY OUTCOMES:
Tumor uptake | 90days
  The standardized uptake value (SUV) of lesions were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoyan Liu, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No